CLINICAL TRIAL: NCT03568565
Title: Web-based Marriage Preparation/Enrichment and Divorce Prevention for Low-Income Couples
Brief Title: Automated & Coached Web-based Programs to Improve and Strengthen Romantic Relationships
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Children's Bureau - Administration for Children and Families (Other)
Responsible Party: Principal Investigator, Brian D Doss, Professor, University of Miami
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 20160451-R
Record Dates: First submitted 2018-06-06; First posted 2018-06-26 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Relationship, Marital

STUDY DESIGN:
Intervention Model Description: The model is a partial/limited SMART design. Couples are initially randomly assigned to one of five groups - a waitlist control, the ePREP program (with and without a coach) and the OurRelationship program (with and without a coach). Following initial randomization, couples initially assigned to complete either program without a coach and who are not completing activities in a timely manner will be re-randomized to either continue without a coach or received a coach.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- ePREP Program (Experimental): The ePREP program is based on the in-person Prevention and Relationship Enhancement Program. The ePREP program consists of six sections of material. In each section, new information and skills are presented, videos demonstrate real couples practicing the skills, participants are encouraged to discuss the information in the context of their own relationship, and a multiple choice quiz reiterates and summarizes the section. In addition to the core educational materials, couples are asked to complete six additional online and offline homework assignments (one per week), each lasting approximately one hour. Participants who do not complete activities in a timely manner will be re-randomized to either continue without a coach or to receive a coach.
  Interventions: Behavioral: ePREP Program
- ePREP Program plus Coach (Experimental): The ePREP program is based on the in-person Prevention and Relationship Enhancement Program. The ePREP program consists of six sections of material. In each section, new information and skills are presented, videos demonstrate real couples practicing the skills, participants are encouraged to discuss the information in the context of their own relationship, and a multiple choice quiz reiterates and summarizes the section. In addition to the core educational materials, couples are asked to complete six additional online and offline homework assignments (one per week), each lasting approximately one hour. Couples also have four, brief video or phone calls with a coach throughout the program.
  Interventions: Behavioral: ePREP Program
- OurRelationship Program (Experimental): The OurRelationship program is based on Integrative Behavioral Couple Therapy and encourages couples to select, understand, and solve a relationship problem. Partners complete the majority of the web-based program on their own and come together for three key conversations with their partner.Participants who do not complete activities in a timely manner will be re-randomized to either continue without a coach or to receive a coach.
  Interventions: Behavioral: OurRelationship Program
- OurRelationship Program plus Coach (Experimental): The OurRelationship program is based on Integrative Behavioral Couple Therapy and encourages couples to select, understand, and solve a relationship problem. Partners complete the majority of the web-based program on their own and come together for three key conversations with their partner. The first conversation between partners centers on discussing possible core relationship issues and jointly deciding on the problem(s) to focus on during the program. During the second conversation, both partners' previous written responses are displayed on the screen and conversation is encouraged. During the final conversation, couples share their strategies to decrease stress, improve patterns of communication, and engage in problem-solving exercises specific to their core issue(s). Couples also have four, brief video or phone calls with a coach throughout the program.
  Interventions: Behavioral: OurRelationship Program
- Waitlist (No Intervention): Participants are assessed at 1, 2, 4, and 6 months after randomization; however, no active intervention is given during the waitlist period.

INTERVENTIONS:
Behavioral: ePREP Program — see arm descriptions
  Arms: ePREP Program; ePREP Program plus Coach
Behavioral: OurRelationship Program — see arm descriptions
  Arms: OurRelationship Program; OurRelationship Program plus Coach

SUMMARY:
This study investigates the effectiveness of self-help, web-based programs to improve romantic relationships and related outcomes. Couples will be randomly assigned to complete the OurRelationship program, the ePREP program, the OurRelationship program with the addition of a coach, the ePREP program with the addition of a coach, or a wait-list control group and followed for six months.

DETAILED DESCRIPTION:
Nationwide, lower-income (LI) couples (those with household incomes <200% of the federal poverty level) - many of whom are also African American, Hispanic/Latino, or rural couples - face numerous challenges to their relationships. Chief amongst those challenges are: 1) higher risk of relationship problems and 2) lack of access to effective relationship services to prevent or intervene with relationship distress. Compared to higher-income couples, LI married and cohabiting couples are significantly more likely to divorce or separate and report lower relationship quality. Unfortunately, LI couples are least likely to receive interventions to prevent or solve relationship problems. To overcome these barriers, we propose to test the effectiveness of two effective web-based curricula - OurRelationship and PREP Online.

A total of 1,246 LI couples will be recruited nationwide and randomly assigned to the ePREP program, the OurRelationship program, the ePREP program plus a coach, the OurRelationship program plus a coach, or a wait-list control group and followed for six months. Once randomly assigned to group, couples will be assessed at one month, two months, four months, and six months following randomization. After couples randomized to the wait-list control group finish their waiting period, they will be able to select the program they would like to complete (OurRelationship or ePREP) but will not complete research assessments during or following their participation in the program.

ELIGIBILITY:
Inclusion Criteria:

1. They are married, engaged, or have been cohabiting with their partner for at least six months
2. They are both located in the United States
3. Both partners are willing to participate in the study
4. Both partners are between the ages of 18 and 64 (inclusive)
5. Couples report a household income at or below 200% of the Federal Poverty Level.

Exclusion Criteria:

1. Severe domestic violence
2. Inadequate internet connection
3. Previous participation in OR, PREP-O, in-person PREP, or its variants
4. Current participation in other relationship programs
5. Current participation in an evaluation funded by Administration for Children and Families

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2500 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Change in Relationship Satisfaction | Baseline, 2 months after baseline, and 6 months after baseline
  Four-item Couple Satisfaction Index (CSI) self-report measure. Range of scores 0 to 21, with higher scores indicating greater satisfaction.

SECONDARY OUTCOMES:
Change in Communication Conflict | Baseline, 2 months after baseline, and 6 months after baseline
  7-item scale; self-report of communication conflict. Range of scores 7 to 28, with higher scores indicating greater conflict.
Relationship break-up potential | Baseline, 2 months after baseline, and 6 months after baseline
  3-item self-report measure of likelihood of relationship ending in the near future. Range of scores 3 to 15, with higher scores indicating greater potential for the relationship to end.

CONTACTS AND LOCATIONS:
Overall Officials: Brian D Doss, Ph.D., Principal Investigator — Professor
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be provided to Administration for Children and Families to facilitate secondary data analyses.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified data provided to ACF within 6 months of study completion. De-identified data available to outside researchers 1.5 years after enrollment ends.
Access Criteria: Available to researchers who have approval from their local IRB.

REFERENCES:
- [Derived] Le Y, Roddy MK, Rothman K, Salivar EG, Guttman S, Doss BD. A randomized controlled trial of the online OurRelationship program with varying levels of coach support. Internet Interv. 2023 Aug 28;34:100661. doi: 10.1016/j.invent.2023.100661. eCollection 2023 Dec. PMID 37674656
- See also: To learn more about the study — http://www.CouplesResearch.com